CLINICAL TRIAL: NCT00476671
Title: Prevalence and Risk Factors of HIV-associated Neurocognitive Impairment and Psychiatric Comorbidities in HIV-1 Infected Thai Individuals With Undetectable Viral Load in the HAART Era.
Brief Title: Neurocognitive Impairment and Psychiatric Comorbidities in HIV-1
Status: Completed | Type: Observational
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: University of Hawaii (Other); SEARCH Research Foundation (Other); Chulalongkorn University (Other); University of Missouri, Department of Psychology, Division of Neuroscience (Other)
Responsible Party: Sponsor
Other Study IDs: HIV-NAT 040
Record Dates: First submitted 2007-05-20; First posted 2007-05-22 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: HIV Infections
Keywords: neuropsychiatric; neurocognitive; psychiatric; HIV related dementia; MCMD; HIV-1; Prevalence, risk factors of neurocognitive impairment and psychiatric comorbidities in HIV-1 infected patients with undetectable viral load in the HAART era.; Treatment Experienced
MeSH Terms: conditions — HIV Infections; AIDS Dementia Complex | interventions — Spinal Puncture; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — PBMC and plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: HIV infected adults with viral load < 50 copies/ml on NNRTI based HAART
  Interventions: Procedure: lumbar puncture, MRI, MRS

INTERVENTIONS:
Procedure: lumbar puncture, MRI, MRS — lumbar puncture, MRI, MRS are only performed in patients with HIV associated dementia

SUMMARY:
To assess the prevalence and risk factors of neurocognitive impairment and psychiatric comorbidities in HIV infected patients who have undetectable viral load, have been on HAART for at least 1 year and have no history of CNS infection.

DETAILED DESCRIPTION:
To understand how to prevent and treat HIV-associated neurocognitive impairment and psychiatric comorbidities in HIV-infected Thai individuals who don't have current AIDS related illness or current and prior central nervous system (CNS) infection, and have been well treated with HAART with undetectable HIV RNA.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Evidence of HIV infection (confirmed positive ELISA and documented history of measurable HIV RNA)
* Age > 18 years old
* Plasma HIV RNA of < 50 copies/ml within 3 months prior to screening
* Have been on only NNRTI-based HAART regimen for the entire duration and for at least1 year.

Exclusion Criteria:

* Current AIDS defining illnesses
* Current or history of previous CNS infection.
* Head injury with loss of consciousness greater than 1 hour
* Acute illness within 30 days prior to entry that, in the opinion of investigators, would prevent patients from completing the protocol required procedures.
* Known learning disability including dyslexia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV infected adults with viral < 50 copies/ml on NNRTI based HAART
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2007-03; Primary Completion 2008-04 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Neuropsychological testing score | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Jintanat Ananworanich, MD, Ph.D, Principal Investigator — The HIV Netherlands Australia Thailand Research Collaboration
Locations (1):
- The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT), Bangkok, Thailand

REFERENCES:
- See also: The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org